CLINICAL TRIAL: NCT02834390
Title: Phase 1b, Open-label, Dose Escalation Study of Quizartinib in Combination With Induction and Consolidation Chemotherapy in Japanese Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: Study of Quizartinib in Japanese Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC220-A-J102
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Results first posted 2021-08-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; phase 1; hematology; malignancy; newly diagnosed
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — quizartinib; Cytarabine; Idarubicin; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Quizartinib 20 mg/day (Experimental): Participants who received 20 mg quizartinib once daily in the morning under fasting conditions.
  For the Induction phase, cytarabine (100 mg/m^2/day IV) and either idarubicin (12 mg/m^2/day IV infusion) or daunorubicin (60 mg/m^2/day IV) were co-administered with quizartinib.
  For the Consolidation phase, cytarabine (3.0 g/m^2/12 hours IV) was co-administered with quizartinib.
  Interventions: Drug: Quizartinib; Drug: Cytarabine; Drug: Idarubicin; Drug: Daunorubicin
- Quizartinib 40 mg/day (Experimental): Participants who received 40 mg quizartinib once daily in the morning under fasting conditions.
  For the Induction phase, cytarabine (100 mg/m^2/day IV) and either idarubicin (12 mg/m^2/day IV infusion) or daunorubicin (60 mg/m^2/day IV) were co-administered with quizartinib.
  For the Consolidation phase, cytarabine (3.0 g/m^2/12 hours IV) was co-administered with quizartinib.
  Interventions: Drug: Quizartinib; Drug: Cytarabine; Drug: Idarubicin; Drug: Daunorubicin

INTERVENTIONS:
Drug: Quizartinib — [Induction period, Cycle 1] Once-daily repeated oral administration Day 8 to Day 21.
  [Induction period, Cycle 2] Once-daily repeated oral administration Day 6 to Day 19.
  [Consolidation period] Once-daily repeated oral administration Day 6 to Day 19.
Drug: Cytarabine — [Induction period, Cycle 1] Once-daily intravenous injection of 100 mg/m^2 cytarabine on Day 1 to 7.
  [Induction period, Cycle 2] Once-daily intravenous injection of 100 mg/m^2 cytarabine on Day 1 to 5.
  [Consolidation period] Twice-daily intravenous injection of 3.0 g/m^2 cytarabine at 12-hour intervals on Days 1, 3, and 5.
Drug: Idarubicin — Either Idarubicin or Daunorubicin will be used [Induction period, Cycle 1] Once-daily intravenous injection of 12 mg/m^2 idarubicin on Day 1 to 3.
  [Induction period, Cycle 2] Once-daily intravenous injection of 12 mg/m^2 idarubicin on Day 1 and 2.
Drug: Daunorubicin — Either Idarubicin or Daunorubicin will be used [Induction period, Cycle 1] Once-daily intravenous injection of 60mg/m^2 daunorubicin on Day 1 to 3.
  [Induction period, Cycle 2] Once-daily intravenous injection of 60mg/m^2 daunorubicin on Day 1 and 2.

SUMMARY:
This is a phase 1b, dose escalation, study of quizartinib to evaluate the safety profile, the pharmacokinetics, and the recommended dose of quizartinib for subsequent clinical studies of the combination of quizartinib and induction and consolidation chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* No prior treatment for AML (including quizartinib)
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0 to 2

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia
* Active acute or chronic systemic fungal, bacterial, or viral infection not well controlled by antifungal, antibacterial or antiviral therapy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-08-12 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 7 participants who met all inclusion and no exclusion criteria were enrolled and received treatment in the study.
Groups:
- Quizartinib 40 mg/Day: Participants who received 40 mg/day quizartinib once daily in the morning under fasting conditions.
  For the Induction phase, cytarabine (100 mg/m^2/day IV) and either idarubicin (12 mg/m^2/day IV infusion) or daunorubicin (60 mg/m^2/day IV) were co-administered with quizartinib.
  For the Consolidation phase, cytarabine (3.0 g/m^2/12 hours IV) was co-administered with quizartinib.
Period: Induction Phase
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day
Started | 4 | 3
Completed | 2 | 1
Not Completed | 2 | 2
Not completed — Progressive disease | 0 | 1
Not completed — CR, CRp, or CRi not achieved (Induction Cycle 2) | 2 | 0
Not completed — Relapse after CR, CRp, or CRi | 0 | 1
Period: Consolidation Phase
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day
Started | 2 | 1
Completed | 1 | 0
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (10.5) | 53.7 (17.1) | 55.9 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Summary of Best Responses After a Daily Dose of 20 mg or 40 mg in Combination With Standard Chemotherapy to Japanese Participants With Newly Diagnosed Acute Myeloid Leukemia (AML)
Description: Best response was defined as the best measured complete remission (CR), CR with incomplete hematological recovery (CRi), CR with incomplete platelet recovery (CRp), Partial remission (PR), or No response (NR) in the overall response assessments at all time points after the first dose. CR is defined as absence of leukemia cells morphologically; bone marrow blasts <5 %; neutrophil count ≥ 1000 /mm 3; platelet count ≥ 100 ,000 /mm 3, independence of RBC transfusions for 4 weeks; independence of platelet transfusions for 1 week; absence of extramedullary leukemia.
Time Frame: Day 0 to Day 21 of last completed cycle (each cycle 28 days), up to approximately 1 year
Population: Best response was assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day
Number analyzed (Participants) | 4 | 3
Participants
  Complete remission (CR) | 0 | 0
  CR with incomplete platelet recovery (CRp) | 0 | 0
  CR with incomplete hematological recovery (CRi) | 3 | 2
  Partial remission (PR) | 1 | 0
  No response (NR) | 0 | 1

2. Primary Outcome: Summary of Best Response Rates After the First Oral Dose of Quizartinib in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: Best response was defined as the best measured complete remission (CR), CR with incomplete hematological recovery (CRi), CR with incomplete platelet recovery (CRp), Partial remission (PR), or No response (NR) in the overall response assessments at all time points after the first dose.
Time Frame: Day 0 to Day 21 of last completed cycle (each cycle 28 days), up to approximately 1 year
Population: Best response was assessed in the Efficacy Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day
Number analyzed (Participants) | 4 | 3
percentage of participants
  Composite CR rate (CRc rate: CR+CRp+CRi) | 75.0 [30.1 to 95.4] | 66.7 [20.8 to 93.9]
  Response rate (CRc+PR) | 100 [51.0 to 100.0] | 66.7 [20.8 to 93.9]

3. Primary Outcome: Pharmacokinetic Parameter Maximum Serum Concentration (Cmax) of Geometric Means of Quizartinib and Active Metabolite (AC886) After Daily Dose of 20 mg or 40 mg Combined With Chemotherapy to Japanese Participants With Newly Diagnosed Acute Myeloid Leukemia
Description: The maximum serum plasma concentration (Cmax) is reported at Induction phase Cycle 1, Day 9 and the maximum serum plasma concentration at steady state (Cmax,ss) is reported at Induction phase Cycle 1, Day 21 for quizartinib, active metabolite AC886, and quizartinib and AC886.
Time Frame: Induction phase Cycle 1, Day 8 to Cycle 1, Day 21 (each cycle 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day
Number analyzed (Participants) | 4 | 3
ng/mL
  Cycle 1, Day 8: Quizartinib, Cmax | 42.4 (25.7) | 91.3 (28.5)
  Cycle 1, Day 8: AC886, Cmax | 36.5 (25.4) | 103 (37.0)
  Cycle 1, Day 8: Quizartinib + AC886, Cmax | 77.4 (10.3) | 180 (16.0)
  Cycle 1, Day 21: Quizartinib, Cmax, ss: number analyzed (Participants) | 4 | 2
  Cycle 1, Day 21: Quizartinib, Cmax, ss | 64.2 (64.0) | 212 (47.4)
  Cycle 1, Day 21: AC886, Cmax, ss: number analyzed (Participants) | 4 | 2
  Cycle 1, Day 21: AC886, Cmax, ss | 96.7 (23.7) | 256 (45.0)
  Cycle 1, Day 21: Quizartinib + AC886, Cmax: number analyzed (Participants) | 4 | 2
  Cycle 1, Day 21: Quizartinib + AC886, Cmax | 162 (35.3) | 480 (2.4)

4. Primary Outcome: Pharmacokinetic Parameter Area Under the Concentration-Time Curve During Dosing Interval of Quizartinib and Metabolite (AC886) After Daily Dose of 20 mg or 40 mg With Chemotherapy to Japanese Participants With Newly Diagnosed Acute Myeloid Leukemia
Description: The area under the plasma concentration-time curve during dosing interval (AUCtau) of geometric means is reported at Induction phase Cycle 1, Day 9 and the area under the plasma concentration-time curve during dosing interval at steady state (AUCtauss) of geometric means are reported at Induction phase Cycle 1, Day 21 for quizartinib, active metabolite AC886, and quizartinib and AC886.
Time Frame: Induction phase Cycle 1, Day 8 to Cycle 1, Day 21 (each cycle 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day
Number analyzed (Participants) | 4 | 3
ng*h/mL
  Cycle 1, Day 8: Quizartinib, AUCtau | 418 (50.4) | 921 (31.3)
  Cycle 1, Day 8: AC886, AUCtau | 555 (28.8) | 1640 (24.4)
  Cycle 1, Day 8: Quizartinib + AC886, AUCtau | 1010 (26.9) | 2640 (8.0)
  Cycle 1, Day 21: Quizartinib, AUCtau,ss: number analyzed (Participants) | 4 | 2
  Cycle 1, Day 21: Quizartinib, AUCtau,ss | 991 (87.7) | 2940 (76.6)
  Cycle 1, Day 21: AC886, AUCtau, ss: number analyzed (Participants) | 4 | 2
  Cycle 1, Day 21: AC886, AUCtau, ss | 1940 (25.4) | 5310 (40.6)
  Cycle 1, Day 21: Quizartinib + AC886, AUCtau: number analyzed (Participants) | 4 | 2
  Cycle 1, Day 21: Quizartinib + AC886, AUCtau | 3020 (42.3) | 8850 (0.3)

5. Primary Outcome: Pharmacokinetic Parameter Time of Maximum Plasma Concentration (Tmax) of Quizartinib and the Active Metabolite (AC886) After a Daily Dose of 20 mg or 40 mg Combined With Chemotherapy to Japanese Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Description: The time of maximum plasma concentration (Tmax) of geometric means is reported at Induction phase Cycle 1, Day 9 and the time of maximum plasma concentration at steady state (Tmax,ss) of geometric means is reported at Induction phase Cycle 1, Day 21 for quizartinib, active metabolite AC886, and quizartinib and AC886.
Time Frame: Induction phase Cycle 1, Day 8 to Cycle 1, Day 21 (each cycle 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hour
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day
Number analyzed (Participants) | 4 | 3
hour
  Cycle 1, Day 8: Quizartinib, Tmax | 3.03 [1.05 to 6.03] | 2.17 [2.07 to 4.17]
  Cycle 1, Day 8: AC886, Tmax | 5.01 [2.05 to 6.03] | 6.08 [4.03 to 6.17]
  Cycle 1, Day 8: Quizartinib + AC886, Tmax | 4.01 [2.05 to 6.03] | 4.17 [4.03 to 6.17]
  Cycle 1, Day 21: Quizartinib, Tmax,ss: number analyzed (Participants) | 4 | 2
  Cycle 1, Day 21: Quizartinib, Tmax,ss | 4.03 [2.03 to 4.13] | 4.08 [4.05 to 4.12]
  Cycle 1, Day 21: AC886, Tmax,ss: number analyzed (Participants) | 4 | 2
  Cycle 1, Day 21: AC886, Tmax,ss | 5.02 [2.08 to 5.98] | 6.09 [6.05 to 6.13]
  Cycle 1, Day 21: Quizartinib + AC886, Tmax: number analyzed (Participants) | 4 | 2
  Cycle 1, Day 21: Quizartinib + AC886, Tmax | 4.03 [2.08 to 5.93] | 4.08 [4.05 to 4.12]

6. Primary Outcome: Pharmacokinetic Parameter Metabolite to Parent Ratio (MR) of Active Metabolite (AC886) After a Daily Dose of 20 mg or 40 mg Combined With Chemotherapy to Japanese Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Description: The metabolite to parent ratio of geometric means for Cmax and AUCtau is reported at Induction phase Cycle 1, Day 9 for active metabolite AC886 is reported.
Time Frame: Induction phase Cycle 1, Day 8 (each cycle 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: metabolite to parent ratio
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day
Number analyzed (Participants) | 4 | 3
metabolite to parent ratio
  Cycle 1, Day 8: MR (Cmax) | 0.861 (43.8) | 1.13 (45.6)
  Cycle 1, Day 8: MR (AUCtau) | 1.33 (64.1) | 1.78 (56.4)

7. Primary Outcome: Pharmacokinetic Parameter Trough Plasma Concentration (Ctrough) of Quizartinib and Active Metabolite (AC886) After a Daily Dose of 20 mg or 40 mg Combined With Chemotherapy to Japanese Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Description: The trough plasma concentration (Ctrough) of geometric means is reported at Induction phase Cycle 1, Day 21 for serum quizartinib, active metabolite AC886, and quizartinib and AC886.
Time Frame: Induction phase Cycle 1, Day 21 (each cycle 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day
Number analyzed (Participants) | 4 | 2
ng/mL
  Cycle 1, Day 21: Quizartinib | 22.7 (173.4) | 77.1 (117.6)
  Cycle 1, Day 21: AC886 | 68.6 (49.3) | 195 (46.1)
  Cycle 1, Day 21: Quizartinib + AC886 | 94.6 (68.5) | 299 (3.3)

8. Primary Outcome: Pharmacokinetic Parameter Accumulation Ratio (AR) of Quizartinib and Active Metabolite (AC886) After a Daily Dose of 20 mg or 40 mg Combined With Chemotherapy to Japanese Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Description: The accumulation ratio of geometric means for Cmax and AUCtau is reported at Induction phase Cycle 1, Day 21 for serum quizartinib, active metabolite AC886, and quizartinib and AC886.
Time Frame: Induction phase Cycle 1, Day 21 (each cycle 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: accumulation ratio
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day
Number analyzed (Participants) | 4 | 2
accumulation ratio
  Cycle 1, Day 21: Quizartinib AR (Cmax) | 1.52 (72.1) | 1.98 (58.5)
  Cycle 1, Day 21: AC886 AR (Cmax) | 2.65 (46.9) | 2.55 (7.2)
  Cycle 1, Day 21: Quizartinib + AC886 AR (Cmax) | 2.09 (41.6) | 2.53 (16.2)
  Cycle 1, Day 21: Quizartinib AR (AUCtau) | 2.37 (88.5) | 2.84 (36.2)
  Cycle 1, Day 21: AC886 AR (AUCtau) | 3.50 (56.2) | 3.31 (5.4)
  Cycle 1, Day 21: Quizartinib + AC886 AR (AUCtau) | 2.99 (59.5) | 3.24 (6.8)

9. Primary Outcome: Number of Participants Treatment-Emergent Adverse Events Reported During Induction Phase After a Daily Dose of 20 mg or 40 mg in Combination With Standard Chemotherapy to Japanese Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event (AE) that emerges (or worsens) from the first dose of study drug and coadministered drugs to the follow-up visit, 35 days after the last dose of study drug and coadministered drugs, or the start date of new AML post-treatment, whichever was earlier.
Time Frame: Induction phase Cycle 1, Day 1 up to 35 days after last dose in Cycle 2 (each cycle 28 days), up to approximately 1 year
Population: Adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day
Number analyzed (Participants) | 4 | 3
Participants
  Participants with TEAEs | 4 | 3
  Infections and Infestations | 1 | 3
  Pneumonia | 1 | 1
  Skin infection | 0 | 1
  Staphylococcal bacteraemia | 0 | 1
  Blood and Lymphatic System Disorders | 4 | 3
  Febrile neutropenia | 4 | 3
  Anaemia | 2 | 1
  Leukopenia | 1 | 0
  Neutropenia | 1 | 0
  Thrombocytopenia | 1 | 0
  Immune Disorders | 0 | 1
  Hypersensitivity | 0 | 1
  Metabolism and Nutrition Disorders | 3 | 2
  Decreased appetite | 3 | 1
  Hypoalbuminaemia | 1 | 1
  Hypokalaemia | 2 | 0
  Hypomagnesaemia | 1 | 0
  Hyponatraemia | 1 | 0
  Hypophosphataemia | 1 | 0
  Hypouricaemia | 0 | 1
  Tumour lysis syndrome | 1 | 0
  Nervous System Disorders | 2 | 1
  Dysgeusia | 2 | 1
  Dizziness | 1 | 0
  Eye Disorders | 1 | 0
  Photophobia | 1 | 0
  Cardiac Disorders | 0 | 1
  Palpitations | 0 | 1
  Vascular Disorders | 0 | 1
  Hypotension | 0 | 1
  Respiratory, Thoracic, and Mediastinal Disorders | 0 | 1
  Epistaxis | 0 | 1
  Oropharyngeal pain | 0 | 1
  Respiratory disorder | 0 | 1
  Gastrointestinal Disorders | 3 | 3
  Abdominal pain upper | 3 | 1
  Nausea | 2 | 2
  Constipation | 1 | 2
  Diarrhoea | 1 | 2
  Stomatitis | 2 | 1
  Cheilitis | 1 | 1
  Vomiting | 1 | 1
  Melaena | 0 | 1
  Hepatobiliary Disorders | 0 | 1
  Hepatic function abnormal | 0 | 1
  Skin and Subcutaneous Tissue Disorders | 4 | 3
  Alopecia | 3 | 2
  Rash | 1 | 2
  Rash maculo-papular | 1 | 1
  Dermatitis bullous | 0 | 1
  Dry skin | 0 | 1
  Musculoskeletal and Connective Tissue Disorders | 1 | 3
  Arthralgia | 0 | 2
  Musculoskeletal pain | 0 | 1
  Myalgia | 1 | 0
  Pain in extremity | 0 | 1
  Renal and Urinary Disorders | 1 | 0
  Haematuria | 1 | 0
  Proteinuria | 1 | 0
  Urinary tract pain | 1 | 0
  Reproductive System and Breast Disorders | 0 | 1
  Menorrhagia | 0 | 1
  General Disorders & Administration Site Conditions | 0 | 1
  Oedema peripheral | 0 | 1
  Pyrexia | 0 | 1
  Investigations | 4 | 3
  Gamma-glutamyltransferase increased | 3 | 1
  Alanine aminotransferase increased | 2 | 1
  Blood alkaline phosphatase increased | 1 | 1
  Electrocardiogram QT prolonged | 0 | 2
  Platelet count decreased | 1 | 1
  Weight decreased | 1 | 1
  White blood cell count decreased | 1 | 1
  Aspartate aminotransferase | 1 | 0
  Aspartate aminotransferase increased | 0 | 1
  Blood bilirubin increased | 1 | 0
  Blood lactate dehydrogenase increased | 0 | 1
  Blood pressure decreased | 0 | 1
  Lipase increased | 0 | 1

10. Primary Outcome: Number of Participants Treatment-Emergent Adverse Events Reported During Consolidation Phase After a Daily Dose of 20 mg or 40 mg in Combination With Standard Chemotherapy to Japanese Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Description: as for outcome 9
Time Frame: Consolidation phase Cycle 1, Day 1 up to 35 days after last dose (each cycle 28 days), up to approximately 1 year
Population: Adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day
Number analyzed (Participants) | 2 | 1
Participants
  Participants with TEAEs | 2 | 1
  Infections and Infestations | 1 | 1
  Lung infection | 0 | 1
  Skin infection | 1 | 0
  Upper respiratory tract infection | 1 | 0
  Blood and Lymphatic System Disorders | 2 | 1
  Febrile neutropenia | 2 | 1
  Nervous System Disorders | 1 | 0
  Dysgeusia | 1 | 0
  Gastrointestinal Disorders | 2 | 0
  Diarrhoea | 2 | 0
  Nausea | 1 | 0
  Stomatitis | 1 | 0
  Skin and Subcutaneous Tissue Disorders | 1 | 1
  Rash | 1 | 0
  Rash maculo-papular | 0 | 1
  General Disorders & Administration Site Conditions | 1 | 0
  Oedema peripheral | 1 | 0
  Investigations | 2 | 1
  Platelet count decreased | 1 | 1
  White blood cell count decreased | 1 | 1
  Alanine aminotransferase increased | 1 | 0
  Electrocardiogram QT prolonged | 0 | 1
  Injury, Poisoning, and Procedural Complications | 0 | 1
  Contusion | 0 | 1
  Fall | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from Induction phase Cycle 1, Day 1 up to 35 days after last completed cycle in Consolidation phase, up to approximately 1 year.
Description: A treatment-emergent AE was defined as an AE that emerges (or worsens) from the first dose of study drug and coadministered drugs to the follow-up visit, 35 days after the last dose of study drug and co-administered drugs, or the start date of new acute myeloid leukemia post-treatment, whichever was earlier. The serious AEs (SAEs) reported occurred only in the Induction phase. No SAEs occurred during the consolidation phase. TEAEs at ≥5% are reported for both induction and consolidation phases.
Arm/Group | Quizartinib 20 mg/Day | Quizartinib 40 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quizartinib 20 mg/Day (N=4) | Quizartinib 40 mg/Day (N=3)
Pneumonia (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quizartinib 20 mg/Day (N=4) | Quizartinib 40 mg/Day (N=3)
Pneumonia (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 3
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Cheilitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 1
Aspartate aminotransferase (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT02834390/Prot_SAP_000.pdf